CLINICAL TRIAL: NCT06204159
Title: Lipiodol Deposition in Hypervascular Tumors: Endhole vs. Pressure-modulated Delivery
Brief Title: Lipiodol Deposition Using Endhole vs. Pressure-Modulated Delivery
Acronym: Trinav
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: TriSalus Life Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UPCC 01223; 853163 (Other: University of Pennsylvania IRB)
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Carcinoma; Neuroendocrine Tumors
Keywords: TACE; Catheter
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neuroendocrine Tumors

STUDY DESIGN:
Intervention Model Description: Exploratory
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- End Hole Catheter followed by TriNav Catheter (Experimental): FDA approved catheter
  Randomization End Hole catheter then TriNav catheter
  Interventions: Device: TACE Catheters
- TriNav Catheter followed by End Hole Catheter (Experimental): FDA approved catheter
  Randomization TriNav catheter then End Hold catheter
  Interventions: Device: TACE Catheters

INTERVENTIONS:
Device: TACE Catheters — End Hole and TriNav catheters are FDA approved. This study is comparing the two for chemotherapy delivery during the TACE procedure.
  This study will randomize which catheter is used for the first TACE procedure and the other catheter will be used for the second TACE procedure

SUMMARY:
The goal of this clinical trial is to compare CT scan of the coverage of tumors treated with TACE using End Hole catheters to those treated with the TriNav catheter that alters tissue pressure. Both catheters are FDA approved for delivery of TACE.

• Is there a difference in CT appearance with delivery in the type of catheter used during the TACE procedure?

Participants will be asked to undergo a TACE procedure, a CT scan and review of their medical record to compare End Hole and TriNav catheters during TACE procedures.

DETAILED DESCRIPTION:
Hepatocellular (HCC) and neuroendocrine (NET) liver metastases undergoing Lipiodol transarterial chemoembolization (TACE) will be randomized to endhole vs. pressure-modulated catheter delivery. Lipiodol deposition will be quantified and correlated with volumetric necrosis, response, and local progression.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged >18 years.
* Plan to undergo lipiodol TACE for HCC or NET liver metastases
* Bilobar disease or distribution for which staged therapy (more than one TACE) for distinct target tumors is planned
* Liver tumor burden does not exceed 50% of the liver volume
* Patent main portal vein
* Life expectancy of greater than 6 months
* ECOG performance status 0-2
* Adequate liver function as measured by: Total bilirubin ≤ 2.0mg/dl, ALT, AST ≤5 times ULN, albumin ≥2.5g/dl
* Adequate marrow and renal function as defined as:
* Platelets >75,000/mcL (may be corrected by transfusion)
* Serum creatinine < 2.0 mg/dl
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such contraception from beginning of study treatment until 1 month following last TACE treatment, as recommended for TACE treatments not conducted within the trial.
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner from first study treatment until 1 month following last TACE treatment.
* Provision of signed and dated informed consent form and ability to consent for oneself.
* Stated willingness to comply with all study procedures and availability for the study duration.

Exclusion Criteria:

* Absolute contraindication to contrast-enhanced MRI
* Absolute contraindication to intravenous iodinated contrast, including history of previous severe contrast reaction or moderate reaction not mitigated by appropriate pre-medication
* Pregnancy or lactation
* Choledochoenteric anastomosis, transpapillary stent or sphincterotomy of duodenal papilla
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
volume and density of lipiodol | immediately following TACE
  To estimate the relative volume and density of lipiodol deposition in hypervascular liver tumors

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pennsylvania, Department of Radiology, Interventional Radiology Division, Philadelphia, Pennsylvania